CLINICAL TRIAL: NCT02494076
Title: Positive Expiratory Pressure for the Treatment of Acute Asthma Exacerbations in Children: A Randomized Controlled Trial
Brief Title: Positive Expiratory Pressure for the Treatment of Acute Asthma in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-1106
Record Dates: First submitted 2014-10-28; First posted 2015-07-10 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Positive-Pressure Respiration; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EzPAP (Experimental): Patients randomized to the EzPAP arm will receive first-line therapies and PEP therapy via EzPAP. All patients will receive 4 cycles with 12 breaths per cycle. 4 cycles is considered one time administration.
  Interventions: Drug: EzPAP
- Standard care (Sham Comparator): Patients randomized to the control arm will receive first-line therapies and standard therapy.
  Interventions: Other: Standard Care

INTERVENTIONS:
Drug: EzPAP
  Other Names: Positive Expiratory Pressure (PEP)
  Arms: EzPAP
Other: Standard Care
  Arms: Standard care

SUMMARY:
Asthma is a leading cause of emergency department (ED) visits for children. A novel way of treating asthma is the use of positive expiratory pressure (PEP). Positive expiratory pressure works by creating pressure in the lungs to keep airways open and to clear mucus from the lungs. PEP is already used in the treatment of asthma at the investigators institution, but studies evaluating the efficacy of PEP therapy in asthma exacerbations do not exist. This study plans to learn more about the use of PEP therapy in the treatment of asthma exacerbations in children in the emergency department. Specifically, the study aims to evaluate if PEP therapy reduces the severity of asthma exacerbations in children and if it reduces the need for additional therapies and admission to the hospital. This study will be a randomized control trial comparing children who receive standard therapy to those who receive standard therapy plus PEP therapy in the treatment of asthma exacerbations. Children age 2 to 18 years presenting to the ED with moderate to severe asthma exacerbations will be included in the study. Reduction in clinical asthma severity will be measured by change in the Pulmonary Asthma Score (the respiratory severity score used at the investigators institution). The need for additional therapies and hospitalization will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 2 and < 18 years of age
* Established diagnosis of asthma, defined as at least two prior episodes of treatment with bronchodilators in their lifetime
* Initial ED presentation with a moderate to severe asthma exacerbation, as defined by a pulmonary asthma score (PAS) >7
* PAS score >7 and <12 after completion of first line therapies (three doses albuterol/ipratropium bromide and oral corticosteroids)

Exclusion Criteria:

* Do not receive complete first line therapies
* Immediately receive a disposition (admission or discharge) as determined by the treating clinician after completion of first line therapies
* Receive prednisone or more than two doses of inhaled bronchodilators prior to main ED evaluation (e.g. during EMS transport or primary care visit)
* Co-morbid illnesses interfering with or contraindicated to usual asthma therapy (e.g. facial or airway abnormalities, pneumonia, chronic lung disease, congenital heart disease, cystic fibrosis, or pneumothorax)
* Critically ill at presentation
* Pregnant women (women known to be pregnant at the time of enrollment)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2017-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nidhya Navanandan, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Navanandan N, Federico M, Mistry RD. Positive Expiratory Pressure for the Treatment of Acute Asthma Exacerbations: A Randomized Controlled Trial. J Pediatr. 2017 Jun;185:149-154.e2. doi: 10.1016/j.jpeds.2017.02.032. Epub 2017 Mar 8. PMID 28284473

RESULTS

PARTICIPANT FLOW:
Groups:
- EzPAP: Patients randomized to the EzPAP arm will receive first-line therapies and PEP therapy via EzPAP. All patients will receive 4 cycles with 12 breaths per cycle.
  EzPAP
- Standard Care: Patients randomized to the control arm will receive first-line therapies and standard therapy.
  Standard Care
Period: Overall Study
Arm/Group | EzPAP | Standard Care
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EzPAP | Standard Care | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 26 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (4.3) | 6.9 (4.1) | 7.8 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 16 | 21 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Asthma Score (PAS)
Description: The primary outcome was the change in asthma severity as determined by change in Pulmonary Asthma Score (PAS) before and after administration of intervention (or control). The same trained, blinded physician assessor, who was not involved in the care of the patient, assessed PAS scores for study subjects before intervention (or control), and 15 minutes after completion of administration. The PAS is a pediatric asthma severity scoring system adapted from previously validated scores, and includes measures of respiratory rate, oxygen saturation, auscultory findings, retractions, and dyspnea. Values from each category are summed producing a total score between 5 and 15. Total scores < 7 correspond with mild asthma exacerbations, while scores ≥ 7 and < 12 indicate moderate asthma, and scores ≥12 to 15 indicate severe asthma. The primary outcome was determined by subtracting the post-intervention score from the pre-intervention score.
Time Frame: 0-30 minutes
Population: 2 patients in EzPAP group were excluded from analysis due to protocol error and missing data.
Measure: Mean (Standard Deviation); unit: mean PAS score
Arm/Group | EzPAP | Standard Care
Number analyzed (Participants) | 24 | 26
mean PAS score | 0.9 (1.2) | 0.4 (1.2)

2. Secondary Outcome: Number of Participants Requiring Second Line Therapies Including Continuous Albuterol, Subcutaneous Terbutaline, IV Magnesium and Supplemental Oxygen After Administration of Intervention or Control
Description: Second line therapies include: continuous albuterol, intravenous magnesium sulfate, subcutaneous or intravenous terbutaline, non-invasive ventilation (BiPAP or CPAP), and supplemental oxygen. The need for these second line therapies will be assessed by the child's treating team in the Emergency Department.
Time Frame: participants will be followed for the duration of ED stay, an expected average of 6-8 hours
Population: 2 subjects excluded from analysis due to missing data
Measure: Count of Participants; unit: Participants
Arm/Group | EzPAP | Standard Care
Number analyzed (Participants) | 24 | 26
Participants
  Continuous albuterol | 11 | 15
  Subcutaneous or intravenous terbutaline | 0 | 1
  Intravenous magnesium | 1 | 3
  Supplemental oxygen | 2 | 7

3. Secondary Outcome: Rate of Inpatient Hospitalization
Description: Number of patients in each group requiring hospital admission
Time Frame: After intervention or control and until follow-up phone call 72 hours after disposition
Population: 2 patients excluded due to missing data and protocol error
Measure: Count of Participants; unit: Participants
Arm/Group | EzPAP | Standard Care
Number analyzed (Participants) | 24 | 26
Participants | 10 | 13

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and collected during the total ED course.
Description: The definition of adverse event does not differ from the clinicaltrials.gov definitions.
Arm/Group | EzPAP | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 3/26 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EzPAP (N=26) | Standard Care (N=26)
Facial redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Light-headedness (Nervous system disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Specific PEP parameters were used that may not have been ideal for the study population. PEP was administered only once. 4 cycles is considered a one time administration. Subsequent administrations were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No